CLINICAL TRIAL: NCT06853080
Title: Feasibility of Using Bortezomib With or Without Chemotherapy in Patients With Atypical Teratoid/Rhabdoid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N202010033
Record Dates: First submitted 2025-02-17; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Atypical Teratoid/Rhabdoid Tumors (AT/RTs); Central Nervous System (CNS) Tumors
MeSH Terms: conditions — Rhabdoid Tumor; Neoplasms | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bortezomib single arm (Experimental): Bortezomib will be administered with chemotherapy on days 1, 4, 8, 11, 22, 25, 29, and 32 of a 56-day treatment cycle for 4 cycles in newly diagnosed patients enrolled on Cohort 1.
  Bortezomib will be administered as a single agent on days 1, 4, 8, 11, 22, 25, 29, and 32 of a 42-day treatment cycle for 4 cycles in all recurrent patients enrolled on Cohort 2.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — 4 cycles of Bortezomib treatment, with each cycle include 8 doses of Bortezomib at 1.3 mg/m2

SUMMARY:
Atypical teratoid/rhabdoid tumors (AT/RTs) account for 1%-2% of all central nervous system (CNS) tumors in children aged 0-14 years, yet are among the most common malignant CNS tumors in infants less than 1 year old. AT/RTs are defined by the loss of INI1 or, rarely, BRG1, encoded by the SMARCB1 and SMARCA4 genes, respectively. Patients with AT/RTs have dismal outcomes due to their highly malignant nature and young age at diagnosis. There remains no standard therapy for AT/RTs. Multimodal treatment strategies include a selective combination of conventional chemotherapy, high dose chemotherapy and stem cell rescue, intrathecal chemotherapy, and radiotherapy after tumor resection. The survival rate, even with aggressive treatment, is still low (2-year survival rate is 32.6%-44.6%). Moreover, currently used cytotoxic therapies incur some neurocognitive side effects, particularly in infants, highlighting the urgent need for novel targeted therapies.

Bortezomib (Velcade®) is the first generation proteasome inhibitor developed by Millennium Pharmaceuticals, Inc. as an anti-cancer medication. Bortezomib was approved by FDA for the treatment of adult patients with multiple myeloma and mantle cell lymphoma (newly diagnosed or relapse/recurrent disease). In children, the safety of BTZ has been proved in phase I clinical trial of patients with acute lymphoblastic leukemia, refractory or recurrent solid tumors, relapsed/refractory high-risk neuroblastoma. Recently, we found the proteasome-encoding genes were highly expressed in AT/RTs compared with that in normal brain tissues, correlated with the malignant phenotype of tumor cells, and were essential for tumor cell survival. Bortezomib targets proteostasis, inhibiting tumor growth and inducing apoptosis through p53 accumulation in three Myc-AT/RT cell lines and in mice with orthotopic xenografts of AT/RT. Our findings suggest that BTZ is a promising targeted therapy for Myc-AT/RTs (manuscript under review). To determine whether the other subgroups of ATRTs (i.e., SHH and TYR subgroups) are sensitive to BTZ, we conducted the in vivo drug test in 2 SHH-AT/RT cell lines (CHLA-02 and CHLA-04). Although CHLA-02 and CHLA-04 cell line were less sensitive to BTZ (IC50 of 15.1 (14.3-15.9) nM and 15.8 (14.5-17.3) nM, respectively) than Myc-AT/RT cell line (IC50 of 5.84 to 8.7 nM), these inhibitory concentrations are still clinically achievable (Cmax, 231.6-312.3 nM). Furthermore, the dependence on ubiquitin proteasome system for survival and high sensitivity to proteasome inhibitors have been reported in SMARCB1-deficient cancer cells. Additionally, we also observed the subgroup shifting in one infant with AT/RTs, from SHH subgroup of primary tumor to Tyr subgroup of the first recurrent tumor and Myc subgroup of the second recurrent tumor. Therefore, we hypothesize that BTZ treatment is potentially effective to all subgroups of CNS AT/RT and propose a clinical trial utilizing BTZ as an add-on therapy to standard and high-dose chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a valid Informed Consent Form signed by the Legal Guardian and/or Patient himself/herself.
2. Patients with CNS AT/RT who were initially diagnosed at the age of 0-20 years.
3. Disease Status:

   Cohort 1: Patients with newly diagnosed AT/RT; Cohort 2: Patients with recurrent or refractory CNS AT/RT who have had at least 1 line of chemotherapy with radiographically measurable disease as defined by at least 1 lesion that can be measured in 2 dimensions.
4. Previous Anticancer Therapy:

   Cohort 1: No previous anticancer chemotherapy other than the use of corticosteroids.

   Cohort 2: Patient has fully recovered from the acute toxic effects of chemotherapy, immunotherapy, or radiation therapy prior to entering this study:
   * Myelosuppressive chemotherapy: Patient has not received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (4 and 6 weeks if prior temozolomide and nitrosourea, respectively).
   * Hematopoietic growth factors: At least 7 days must have elapsed since the completion of therapy with a growth factor. At least 14 days must have elapsed after receiving pegfilgrastim.
   * Biologic (anti-neoplastic agent): At least 7 days must have elapsed since completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur.
   * Monoclonal antibodies: At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody.
   * Radiation therapy: at least 3 months must have elapsed since any irradiation unless measurable disease progression occurs at a site separate from the irradiated area and the patient has recovered from toxicities associated with radiation therapy.
5. Patients must have adequate organ and marrow function as defined below at enrollment and on day 1 of (or within 1 week prior to) each cycle:

   * Absolute Neutrophil Count (ANC) ≥ 1,000/μL
   * Platelets ≥ 100,000/μL at enrollment and on day 1 of each cycle
   * Hemoglobin ≥ 8 g/dL (RBC transfusions allowed)
   * Total bilirubin ≤ 1.5 times institutional upper limit of normal
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 times institutional upper limit of normal (4x ULN if liver involvement)
   * Creatinine ≤ upper limits by age 0-5 years old: 0.8 mg/dL; 6-9 years old: 1.0 mg/dL; 10-12 years old: 1.2 mg/dL; 13-15 years old: male, 1.5 mg/dL; female, 1.4 mg/dL; 16 years or older: male, 1.7 mg/dL; female, 1.4 mg/dL
6. LV Ejection Fraction of ≥ 50% by Echocardiogram
7. Patient must have the Performance status defined by Lansky (< 16 years of age) or Karnofsky (≥16 years of age) Performace Status of ≥ 30 (Cohort 1) or ≥ 60 (Cohort 2).
8. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered to be ambulatory for the purpose of assessing the performance score.
9. Female patients who are at least 10-years-old or are post-menarchal must have a negative serum or urine pregnancy test prior to enrollment
10. Fertile patients must use effective contraception
11. Life expectancy > 8 weeks
12. No evidence of dyspnea at rest
13. Fertile patients must use effective contraception

Exclusion Criteria:

1. Clinically significant medical disorders that could compromise the ability to tolerate protocol therapy or that would interfere with the study procedures or results history.
2. Presence of an active, uncontrolled infection.
3. Existing peripheral neuropathy of NCI CTCAE v5.0 grade 2 or higher.
4. Patients who have not recovered to baseline from previous treatment.
5. Patients with hypersensitivity (not including local reactions) to BTZ, boron, or mannitol.
6. Patients who have been previously treated with BTZ.
7. Requirement for constant administration of strong CYP3A4 interfering agents.
8. Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or with rifampin, rifabutin, rifapentine, or St. John's wort within 7 days prior to initiation of BTZ.
9. Inability to comply with the safety monitoring requirements of the study, as judged by the investigator.
10. Female participants of childbearing potential cannot be pregnant or breast-feeding.
11. Patients who are receiving other investigational drugs 14 or fewer days before enrollment.
12. Patients with extra-CNS, extrarenal rhabdoid tumors or malignant renal rhabdoid tumors without CNS AT/RT are not eligible.
13. Myocardial infarction within 6 months prior to enrollment or New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. If for some reason an electrocardiogram is obtained before study enrollment, any abnormalities detected should be documented as clinically irrelevant.
14. Other severe acute or chronic medical or psychiatric condition or any laboratory abnormality that may increase the risk associated with study participation or investigational product administration or that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
15. Subjects with known active infections requiring ongoing treatment (bacterial, fungal, or viral, including human immunodeficiency virus [HIV]).

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | through study completion, an average of 1 year
  Overall Response Rate (ORR) to bortezomib in patients with recurrent or refractory CNS AT/RT.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | through study completion, an average of 1 year
  Progression-Free Survival (PFS) in patients with newly diagnosed CNS AT/RT
Overall Survival (OS) | through study completion, an average of 1 year
  Overall Survival (OS) in patients with newly diagnosed CNS AT/RT

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Trial still conducted.